CLINICAL TRIAL: NCT01882764
Title: A Phase III Double Blind, Multi-Center Placebo Controlled Maintenance Trial of HMPL-004 in Subjects With Mild to Moderate Ulcerative Colitis With Clinical Remission or Response From Induction Therapy. (NATRUL-4)
Brief Title: HMPL-004 Maintenance Treatment in Subjects With Mild to Moderate Ulcerative Colitis
Acronym: NATRUL-4
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility interim analysis of the Induction Study HMPL-004-03.
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Nutrition Science Partners Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMPL-004-04
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Andrographis paniculata extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HMPL-004 1800 mg/day (Experimental): Subjects qualifying for entry into the Maintenance Phase of the study were randomized to take an oral dose of HMPL-004 (600 mg TID; total dose 1800 mg/day) daily, for 52 weeks.
  Those subjects who demonstrated clinical remission or response after completing the HMPL-004-03 Induction Study, or after completing the Open Label Phase of this study, were eligible for enrollment in the Maintenance Phase of this study.
  Interventions: Drug: HMPL-004
- Placebo (Placebo Comparator): Subjects qualifying for entry into the Maintenance Phase of the study were randomized to take an oral dose of Placebo tablets TID, daily, for 52 weeks.
  Those subjects who demonstrated clinical remission or response after completing the HMPL-004-03 Induction Study, or after completing the Open Label Phase of this study, were eligible for enrollment in the Maintenance Phase of this study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMPL-004 — Remitters and responders from HMPL-004 Induction study and patients complete the 8-week Open Label Induction Phase will be given HMPL-004 orally three times per day with total daily dose of 1800 mg for 52 weeks.
  Other Names: Chuan xinlian
  Arms: HMPL-004 1800 mg/day
Drug: Placebo — Remitters and responders from HMPL-004 Induction study and patients complete the 8-week Open Label Induction Phase will be given Placebo orally three times per day with total daily dose of 1800 mg for 52 weeks.
  Arms: Placebo

SUMMARY:
A study with an 8 week open label phase study followed by a year long placebo controlled maintenance phase in subjects with active mild to moderate ulcerative colitis (UC), with a modified Mayo Score 4-10 and an endoscopy subscore of 2-3, taking mesalamine (or equivalent) as a concomitant medication. Subjects are required to be in clinical remission or clinical response to enter the year long maintenance phase. This study will help evaluate if HMPL-004 is effective in subjects maintaining clinical remission following successful induction therapy achieving clinical remission or clinical response.

DETAILED DESCRIPTION:
A two-phase multi-center study with an open label 8-week induction phase and a randomized, double-blind, placebo controlled maintenance phase to evaluate the efficacy and safety of HMPL-004 for a 52-week maintenance therapy in adults with mild to moderate UC and who have demonstrated a sub-optimal response to mesalamine treatment. The study participants will consist of subjects who have completed either the HMPL-004-03 or HMPL-004-05 induction study, complemented by the enrollment of additional subjects in the open label induction phase who meet the entry criteria of this study. . Subjects entering this maintenance study from one of the HMPL-004 induction studies will have their modified Mayo baseline score from that study as their baseline score for this study. All subjects enrolled in the open label induction phase of the study will be re-evaluated for clinical response and remission after the 8-week open label 2400 mg HMPL-004 treatment period. Clinical responders and remitters will be randomized 2:1 (HMPL-004: placebo) to HMPL-004 1800 mg/day or placebo group for the 52-week maintenance phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of induction study HMPL-004-03 or HMPL-004-05 and achieving clinical remission or response with no disruption of study treatment in the transition to HMPL-004-04, or, for the open label induction phase of the study: have active mild to moderate Ulcerative Colitis defined by a modified Mayo Score of 4 to 10 and with endoscopy score activity of 2-3 points confirmed by a full colonoscopy within 2 weeks prior to study.
2. Subjects must be currently receiving mesalamine ≥ 2.4 g/day (or the equivalent) for at least 6 weeks prior to randomization and on a stable dosage for at least 2 weeks prior to entering the screening phase of the study to ensure a stable dose is established at least 2 weeks prior to the endoscopic procedures.
3. Have adequate renal, hepatic and bone marrow function (see exclusion criteria).
4. Age ≥ 18 years
5. All fertile male and female subjects must agree to use one of the following types of contraception: intrauterine device, implantable progesterone device, progesterone intramuscular injection, oral contraceptive which has been started at least one month prior to visit one and continues for the duration of the trial, contraceptive patch, or condom with spermicide.
6. Show evidence of a personally signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

1. Subjects with intolerance to mesalamine (or equivalent medications).
2. Diagnosed with Crohn's disease or with lesions such as fistulas or granulomas on biopsy noted either in history or at baseline endoscope, which would be suspicious for Crohn's disease, or with a diagnosis of indeterminate colitis.
3. Severe disease with a Ulcerative Colitis modified Mayo Clinic score above 10 points at baseline.
4. Positive stool test for pathogens on sample taken within the 2 weeks prior to study entry.
5. Active clostridium difficile (C. diff) infection.
6. Use of Inflammatory Bowel Disease related herbal supplements including supplements containing andrographis or the use of probiotics two weeks prior to study entry or during the study.
7. Toxic megacolon or toxic colitis.
8. Probable requirement for intestinal surgery within 12 weeks after the start of investigational product.
9. Receiving oral or rectal steroids within 1 month prior to study entry.
10. Receiving rectal mesalamine within 1 week prior to study entry.
11. Receiving azathioprine, 6-mercaptopurine, methotrexate, tacrolimus, cyclosporine, or other immunosuppressive therapy at the time of screening or within the preceding 6 weeks.
12. Receiving anti-tumor necrosis factor-α (TNF-α)agents such as infliximab, adalimumab, golimumab, or certolizumab pegol at the time of screening or within the preceding 8 weeks.
13. Receiving other investigational drugs or biologics within 1 month or five half-lives, whichever is longer.
14. Receiving antibiotics within 2 weeks of study entry.
15. Hemoglobin concentration <9 g/dl.
16. White blood cell count (WBC) below 3,000/cm3, or platelets below 100,000/cm3.
17. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and/or alkaline phosphatase >2.5 upper limit of normal.
18. Serum creatinine >1.5 times upper limit of normal.
19. Significant concurrent medical diseases including: active peptic ulcer disease; uncompensated congestive heart disease; myocardial infarction within the last 12 months; unstable angina pectoris; uncontrolled hypertension; and pulmonary disease requiring oxygen therapy.
20. Chronic Hepatitis B or any history of Hepatitis C.
21. Previous colonic surgery except for simple polypectomy.
22. History of cancer within the last 5 years other than resected cutaneous basal and squamous cell carcinomas, and/or in situ cervical cancer.
23. Subjects with a history of or concurrent colonic dysplasia associated with UC, except those with completely excised sporadic colorectal polyps.
24. Women who are pregnant or breast feeding.
25. Subjects known to be seropositive for HIV, or who have had an AIDS defining illness, or a known immunodeficiency disorder.
26. History of alcohol or drug abuse that would interfere with the ability to be compliant with the study procedure.
27. Known allergy to plants of the Acanthaceae family.
28. Unwillingness to participate in the study.
29. Any underlying medical condition that in the Investigator's opinion will make the administration of study drug hazardous to the subject or would obscure the interpretation of Adverse Events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liu Rongjun, Dr., Study Director — Hutchison Medipharma Limited
Locations (1):
- Clinical Research Management, Inc., Agawam, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HMPL-004 1800 mg/Day | Placebo
Started | 47 | 19
Completed | 0 | 1
Not Completed | 47 | 18

BASELINE CHARACTERISTICS:
Groups:
- HMPL-004 1800 mg/Day: Subjects qualifying for entry into the Maintenance Phase of the study were randomized to take an oral dose of HMPL-004 (600 mg TID; total dose 1800 mg/day) daily, for 52 weeks.
  Those subjects who demonstrated clinical remission or response after completing the HMPL-004-03 Induction Study, or after completing the Open Label Phase of this study, were eligible for enrollment in the Maintenance Phase of this study.
  HMPL-004: Remitters and responders from HMPL-004 Induction study and patients complete the 8-week Open Label Induction Phase will be given HMPL-004 orally three times per day with total daily dose of 1800 mg for 52 weeks.
- Placebo: Subjects qualifying for entry into the Maintenance Phase of the study were randomized to take an oral dose of Placebo tablets TID, daily, for 52 weeks.
  Those subjects who demonstrated clinical remission or response after completing the HMPL-004-03 Induction Study, or after completing the Open Label Phase of this study, were eligible for enrollment in the Maintenance Phase of this study.
  Placebo: Remitters and responders from HMPL-004 Induction study and patients complete the 8-week Open Label Induction Phase will be given Placebo orally three times per day with total daily dose of 1800 mg for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | HMPL-004 1800 mg/Day | Placebo | Total
Number analyzed (Participants) | 46 | 19 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (14.01) | 47.8 (15.64) | 43.4 (14.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 7 | 28
  Male | 25 | 12 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 41 | 16 | 57
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 18 | 56
  Lithuania | 2 | 0 | 2
  Latvia | 1 | 0 | 1
  Bulgaria | 2 | 1 | 3
  Poland | 2 | 0 | 2
  Czechia | 1 | 0 | 1
Current Smoker: Yes, No [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 4
  No | 43 | 18 | 61
Race [Count of Participants; unit: Participants]
  White | 41 | 18 | 59
  Black | 2 | 1 | 3
  Other | 2 | 0 | 2
  Asian | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] | 80.65 (16.70) | 85.99 (24.29) | 82.21 (19.18)
Height [Mean (Standard Deviation); unit: cm] | 170.87 (9.64) | 173.33 (7.99) | 171.59 (9.20)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Achieving Clinical Remission
Description: Clinical remission is defined as a modified Mayo Score ≤2 along with no individual score >1 AND rectal bleeding score = 0.
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 1800 mg/Day | Placebo
Number analyzed (Participants) | 46 | 19
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 56 weeks
Arm/Group | HMPL-004 1800 mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/19
Other Adverse Events (participants affected / at risk) | 11/46 | 4/19
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HMPL-004 1800 mg/Day (N=46) | Placebo (N=19)
Urinary tract infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 2 | 0
URTI (Infections and infestations) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No